CLINICAL TRIAL: NCT00488358
Title: Hemodynamic Changes After Aortic Aneurysm Treatment With Stent-Graft
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01645
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal; aortic; aneurysm; Zenith; blood pressure
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the aortic pulse profile before and after stent-graft implantation to prove that endovascular AAA repair using non-compliant stent-graft changes the aortic pulse profile.

DETAILED DESCRIPTION:
This study will assess hemodynamic changes in aortas of patients after treatment of their abdominal aortic aneurysm (AAA) with an FDA approved stent-graft (Zenith). This study does not require any change in clinical protocol to the the way the AAA procedures are currently done. Utilizing the catheters already employed in this procedure, intravascular blood pressure measurements will be documented at various times and at various anatomic levels prior to and after deployment of the stent-graft.

As the compliant aortic aneurysm acts as a capacitor, expanding during systole and contracting during diastole, it is our hypothesis that endovascular AAA repair using a non-compliant stent-graft changes the aortic pulse profile.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal Aortic Aneurysm with planned treatment using Zenith Endovascular Stent-Graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Abdominal Aortic Aneurysm with planned treatment using Zenith Endovascular Stent-Graft
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2010-01 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jade S Hiramoto, MD, Principal Investigator — Assistant Professor in Residence
Locations (1):
- Division of Vascular Surgery, UCSF, San Francisco, California, United States